CLINICAL TRIAL: NCT05104008
Title: Effectiveness of Lateral Wedge Insole on Knee Osteoarthritis Outcomes in Pakistani Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Rabbiya Riaz, Physiotherapist, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIHS-RABBIYA/Lecturer DPT
Record Dates: First submitted 2021-10-26; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Medial Compartment Knee Osteoarthritis
Keywords: Knee osteoarthritis, functional independence, musculoskeletal physiotherapy, orthotics, quality of life.
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral wedge insoles with home exercises group(Group 1) (Active Comparator): In this group, participants were advised to use lateral wedge insole during walking and long-standing. Non customized full-length lateral wedge insoles of 7mm made of silicon material with 5 degrees angulation (because greater wedging is associated with foot discomfort) was used. Full-length wedge extends under the lesser metatarsal heads which increases the lever arm for rearfoot eversion and thus can prevent subtalar joint rotation. The evaluations were performed every week till fourth week.
  Interventions: Other: Lateral wedge insoles with home exercises group(Group 1)
- Traditional physiotherapy with home exercises group (Group 2) (Active Comparator): Each participant received 40-45 minutes long session, started in lying position. The therapeutic low-intensity pulsed ultrasound (US) was used for 7 minutes with the frequency of 1 MHz, Spatial Average Intensity was 0.2 W /cm2, pulsed duty cycle 20%, therapeutic dose was 112.5 J/cm2 with fixed application on the medial side of the knee joint. The model of US was Unit Intelect Mobile, (Chattanooga Inc). After US therapy passive stretching of calf, hamstring, quadriceps, hip flexors, adductors & abductor s was done, which was followed by the manual strengthening exercises and strengthening with quadriceps bench. The session was repeated thrice a week and 12 sessions per month. The home program was guided in both groups including avoiding low sitting, cross leg sitting along with Isometrics of quadriceps atleast 3 times a day, with 5-10 seconds hold of each contraction.
  Interventions: Other: Traditional physiotherapy with home exercises group (Group 2)

INTERVENTIONS:
Other: Lateral wedge insoles with home exercises group(Group 1) — In this group, participants were advised to use lateral wedge insole during walking and long-standing. Non customized full-length lateral wedge insoles of 7mm made of silicon material with 5 degrees angulation (because greater wedging is associated with foot discomfort) was used. Full-length wedge extends under the lesser metatarsal heads which increases the lever arm for rearfoot eversion and thus can prevent subtalar joint rotation. The evaluations were performed every week till fourth week.
  Arms: Lateral wedge insoles with home exercises group(Group 1)
Other: Traditional physiotherapy with home exercises group (Group 2) — Each participant received 40-45 minutes long session, started in lying position. The therapeutic low-intensity pulsed ultrasound (US) was used for 7 minutes with the frequency of 1 MHz, Spatial Average Intensity was 0.2 W /cm2, pulsed duty cycle 20%, therapeutic dose was 112.5 J/cm2 with fixed application on the medial side of the knee joint. The model of US was Unit Intelect Mobile, (Chattanooga Inc). After US therapy passive stretching of calf, hamstring, quadriceps, hip flexors, adductors & abductor s was done, which was followed by the manual strengthening exercises and strengthening with quadriceps bench. The session was repeated thrice a week and 12 sessions per month. The home program was guided in both groups including avoiding low sitting, cross leg sitting along with Isometrics of quadriceps atleast 3 times a day, with 5-10 seconds hold of each contraction.
  Arms: Traditional physiotherapy with home exercises group (Group 2)

SUMMARY:
Osteoarthritis (OA) is a persistent joint disorder, which normally affects the weight bearing joints especially knee joint. Lateral wedge insole is one such approach suggested by professionals to manage the knee osteoarthritis.Effectiveness of lateral wedge insoles (LWI) group (n=20), and conventional physical therapy (CPT) group (n=20) with home exercises as baseline treatment were assessed on Urdu version of Knee Injury and Osteoarthritis Outcome Score scale (KOOS).

DETAILED DESCRIPTION:
A total of n=104 patients were recruited through the non-probability convenience sampling technique and were thus evaluated for the inclusion criteria. Of which, n=40 participants fulfilled the inclusion criteria. Participants were randomly divided through the sealed envelope method in two groups; lateral wedge insoles with home exercises group (n=20), and traditional physiotherapy with home exercises group (n=20). The data was collected through a general demographic questionnaire and Knee injury and Osteoarthritis Outcome Score (KOOS) in Urdu to determine the severity of pain, stiffness, functional activities, recreational activities and Quality of life to promote functional independence in osteoarthritic patients.[20] The level of significance was set at p<0.05. Statistical Package for the Social Sciences (SPSS) ver. 23 was used for data analysis.As the assumption of the parametric test was met, mixed ANOVA was used for the interaction effect of between-subject factor (group) and within-subject factor (time). With-in group analysis and one way ANOVA was used for between-group comparisons to determine the effect size (ɳp2).

ELIGIBILITY:
Inclusion Criteria:

* Patients with the age criteria of 40-70 years, and who had a history of knee OA were included in the study.

Exclusion Criteria:

* Patients had knee OA due to trauma or any pathology, multiple fractures, or had a medical condition due to which rehabilitation wasn't possible, and not willing to participate in the clinical trials were excluded from the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Knee injury and osteoarthritis outcome pain score | Upto 4 weeks
  Pain associated with daily tasks is measured through Knee injury and osteoarthritis outcome pain score with categories as 'None' for no pain and 'Extreme' for maximum pain value.
Knee injury and osteoarthritis outcome stiffness score | Upto 4 weeks
  It is measured through Knee injury and osteoarthritis outcome stiffness score with categories as 'None' for no stiffness and 'Extreme' for maximum stiffness.
Knee injury and osteoarthritis outcome functional status score | Upto 4 weeks
  Degree of difficulty in performing daily tasks associated with knee joint is measured through Knee injury and osteoarthritis outcome functional status score with categories as 'None' for no difficulty in tasks and 'Extreme' for maximum difficulty in performing tasks. .
Knee injury and osteoarthritis outcome quality of life score | Upto 4 weeks
  Quality of life regarding knee joint disease is measured through Knee injury and osteoarthritis outcome quality of life score with categories as according to patient's satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabbiya Riaz, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR